CLINICAL TRIAL: NCT06465550
Title: A Phase 1 Clinical Trail of the Safety and Efficacy of Gene-modified Autologous Hematopoietic Stem Cell (BD211) Intravenous Infusion for the Treatment of Transfusion-dependent β-thalassaemia Patients
Brief Title: A Phase 1 Study of Gene-modified Autologous Hematopoietic Stem Cell (BD211) Treating β-thalassemia Major
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-TDT-211005
Record Dates: First submitted 2024-06-12; First posted 2024-06-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: β-thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD211 Single-Dose group (Experimental): Route of Administrate: infusion intravenously. Dosage form: injection solution. Dose: ≥ 5×10^6 cells /kg. Frequency of administration: One dosing intravenously. Intervention: Single dose of BD211
  Interventions: Genetic: BD211

INTERVENTIONS:
Genetic: BD211 — Genetically modified CD34+ autologous stem cells were transfused intravenously with single dosing.

SUMMARY:
This study will be intented to evaluate the safety, tolerability, and engraftment efficacy after myeloablative preconditioning and transplantation of autologous CD34+ hematopoietic stem cells transduced with a lentiviral vector encoding the human βA-T87Q-globin gene in patients with transfusion-dependent (TDT) β-thalassemia.

DETAILED DESCRIPTION:
This is an open-label, single-dose study of BD211 in patients with transfusion-dependent β-thalassemia aged 3 to 35 years. It is estimated that 9 subjects will be enrolled. BD211 is a gene modified gene therapy product designed to produce healthy β-globin in red blood cells in beta-thalassemia patients. The total follow-up duration was 18 months, the safe endpoints and effectiveness endpoints will be used to assess the safety and efficacy profiles in patients with transfusion-dependent β-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 3 years (inclusive) to 18 years (exclusive), with no gender restrictions.
2. Parents/legal guardians have fully understood and voluntarily signed a written informed consent form; and it is recommended that children aged 8 and above be involved in the decision to participate in this clinical trial and obtain a written consent form.
3. Transfusion-dependent β-thalassemia patients. "Transfusion-dependent" is defined as: requiring at least 100 mL/kg of packed red blood cells annually; the genotype can be β0/β0, β0/β+, or β+/β+, diagnosed through hemoglobin studies.
4. Eligible for allogeneic hematopoietic stem cell transplantation, but without a donor or those refusing to undergo allogeneic hematopoietic stem cell transplantation.
5. Have undergone symptomatic treatment for at least the past 2 years and have retained medical records including transfusion history.
6. Stable condition and maintained an appropriate iron chelation regimen.
7. Good status of organ function.
8. Good compliance from the individual and parents/legal guardians, willing to adhere to visit schedules, trial plans, laboratory tests, and other trial procedures as stipulated in this protocol.
9. Willing to participate in long-term follow-up research.

Exclusion Criteria:

1. Has a fully HLA-matched hematopoietic stem cell donor and is willing to receive a fully HLA-matched hematopoietic stem cell transplant. Enrollment is otherwise only advised after review by the safety review committee.
2. Positive for antibodies against Human Immunodeficiency Virus 1/2 (HIV-1/HIV-2), Treponema pallidum (TP) specific antibodies, Human T-lymphotropic Virus 1 or 2 (HTLV-1/HTLV-2) antibodies, and Vesicular Stomatitis Virus G (VSV-G).
3. Positive for Hepatitis B Virus (HBV) HbsAg or HBV-DNA; Hepatitis C Virus (HCV) HCAb positive; positive nucleic acid test for Epstein-Barr Virus (EBV) or Cytomegalovirus (CMV).
4. Severe active bacterial, viral, fungal, malarial, or parasitic infections.
5. Has had, or currently has, a malignant, myeloproliferative, or immunodeficiency disorder.
6. Direct relatives with known or suspected hereditary cancer syndromes (including but not limited to breast cancer, colorectal cancer, ovarian cancer, prostate cancer, and pancreatic cancer).
7. Autoimmune diseases that could result in transfusion difficulties.
8. Major organ diseases or abnormal lab tests, including:

   1. Liver cirrhosis, fibrosis, or active hepatitis, and/or abnormal liver function tests (Serum total bilirubin (TBIL) ≥ 1.5x Upper Limit of Normal (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≥ 2.5x ULN; Alkaline phosphatase ≥ 2.5x ULN).
   2. Heart disease, or Left Ventricular Ejection Fraction (LVEF) < 60%.
   3. Kidney diseases, or serum creatinine ≥ 1.5ULN, creatinine clearance rate < 30% of the normal level (measured or calculated by the Cockcroft-Gault equation).
   4. Endocrine disorders, such as insulin-dependent diabetes, hyperthyroidism, or hypothyroidism.
   5. Severe iron overload, serum ferritin ≥ 5000 ng/mL.
   6. Cardiac T2* < 20 ms, and/or liver iron content (LIC) ≥ 15mg/g liver weight by MRI.
   7. Significant pulmonary hypertension diagnosed clinically according to guidelines, requiring clinical medical intervention.
9. Uncorrected bleeding disorders.
10. Severe psychiatric disorders.
11. Peripheral blood white cell (WBC) count < 3x10^9/L or platelets count < 120x10^9/L.
12. Received hydroxyurea treatment within the last 3 months before stem cell collection.
13. Used erythropoiesis-stimulating agents within the 3 months prior to HSC collection.
14. History of allogeneic transplantation.
15. Previously received any type of gene and/or cell therapy.
16. Participating in another clinical trial and is within a 30-day screening period.
17. Has contraindications to anesthesia.
18. Has contraindications to hematopoietic stem cell collection.
19. Allergic to the investigational drug or its excipients.
20. Any other conditions determined by the investigator as unsuitable for participation in this clinical trial.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean time from BD211 treatment to successful neutrophil engraftment, as well as the number and percentage of participants with successful neutrophil engraftment. | 18 months
  Definition of successful neutrophil engraftment: A consistent absolute neutrophil count (ANC) recovery of ≥0.5×10^9/L over three consecutive days.
Mean time from BD211 treatment to successful platelet engraftment, as well as the number and percentage of participants with successful platelet engraftment. | 18 months
  Definition of successful platelet engraftment: No platelet transfusion for 7 days with platelet counts of ≥20×10^9/L in three consecutive measurements.
Proportion of participants achieving transfusion independence (TI) | 18 months
  TI defined as "hemoglobin (Hb) ≥ 90g/L without any transfusion of packed red blood cells (pRBCs) for 12 months at any time during the study period after BD211 treatment"; proportion of participants with TI = number of participants with TI ÷ total number of BD211 treatment.

SECONDARY OUTCOMES:
BD211 transplant-related mortality (TRM) and overall survival (OS) after BD211 treatment. | 18 months
  TRM = number of BD211 transplant-related deaths ÷ total number of BD211 treatment x 100% OS = number of all-cause deaths after BD211 treatment ÷ total number of BD211 treatment x 100%
Incidence of aberrant replication competent lentivirus (RCL) or malignant transformation induced by vector insertion after BD211 treatment. | 18 months
  RCL positivity rate = number of RCL positive cases ÷ total number of BD211 treatment × 100%.
Total number of days hospitalized from the discharge day from LAFR to 18 months after BD211 administration | 18 months
  The number of days of all-cause hospitalisation was calculated for each participant from the start of discharge from the transplantation unit after successful neutrophil and platelet engraftment to 18 months after BD211 treatment .
Types, numbers and incidence rate of adverse events (AEs) and serious adverse events (SAEs) that occurred within 18 months after BD211 adminstration. | 18 months
  AEs and SAEs were evaluated per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.The frequency, severity, and correlation of AEs and SAEs with the investigational drug based on laboratory results and clinical manifestations were determined.
Mean duration (days) after participants reached TI | 18 months
  Mean duration after reaching TI = sum of duration after reaching TI for all participants ÷ total number of participants.
Mean time required from BD211 treatment (D0) to achieve TI | 18 months
  Mean time required from BD211 treatment (D0) to achieve TI = sum of time required from BD211 infusion (D0) to achieve TI ÷ total number of participants.
Mean Hb values after BD211 treatment | 12 months~18months
  Mean Hb of participants per month = sum of Hb (g/L) values of all participants per month ÷ total number of participants
Proportion of participants with 60% and 80% reduction in blood transfusions from baseline | 12 months~18months
  The mean blood transfusion volume (mL/kg/year) in the 2 years prior to enrolment was used as the baseline, and compared with the mean blood transfusion volume (mL/kg/year) in the M12~M18 period after receiving the BD211 infusion, and the proportion of participants whose blood transfusion volume was reduced by 60% and 80%, respectively, was calculated.
Change in ferritin levels from baseline. | 18 months
  Change in mean serum ferritin levels compared to baseline values at 6 months, 12 months and 18 months after BD211 treatment.
Expression of βA-T87Q globin protein in whole blood | 18 months
  HPLC method was used to measure the expression of βA-T87Q globin protein in peripheral blood.
Mean VCN of the BD211 lentivirus vector in peripheral blood | 18 months
  qPCR method were used to measure the VCN level of the BD211 lentivirus vector in peripheral blood.
Dose-response relationship | 18 months
  The relationship between the BD211 dose and efficacy endpoints including TI outcome and expressed level of βA-T87Q globin protein (primarily PD biomarker) in blood were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Sujiang Zhang, M.D., Principal Investigator — Shanghai Ruijin Hospital, Shanghai Jiaotong University; Jianpei Fang, M.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guandong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Shanghai Ruijin Hospital, Shanghai Jiaotong University, Shanghai, Shanghai City